CLINICAL TRIAL: NCT02972645
Title: A First-in-Human, Single Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of LY3305677 in Healthy Subjects
Brief Title: A Study of LY3305677 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Basic Science
Other Study IDs: 16350; I8P-MC-OXAA (Other: Eli Lilly and Company)
Record Dates: First submitted 2016-11-21; First posted 2016-11-23 (Estimated); Last update posted 2017-07-24 (Actual); Status verified 2017-07

CONDITIONS: Healthy
MeSH Terms: interventions — mazdutide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- LY3305677 (Experimental): Single escalating doses of LY3305677 administered subcutaneously (SC)
  Interventions: Drug: LY3305677
- Placebo (Placebo Comparator): Placebo administered SC
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LY3305677 — Administered SC
  Arms: LY3305677
Drug: Placebo — Administered SC
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety of LY3305677 and any side effects that might be associated with it.

This study will also look at how much LY3305677 gets into the blood stream, how long it takes the body to remove it.

This study involves a single dose of LY3305677 administered by subcutaneous injection (SC).

Participation in this study is expected to last up to 16 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Overtly healthy as determined by medical history and physical examination
* Male participants: will agree to use a reliable method of birth control and will not donate sperm during the study and for at least 3 months following the last dose of the investigational product
* Female participants: women not of child-bearing potential due to surgical sterilization confirmed by medical history or menopause
* First generation Japanese participants or non-Japanese participants
* Have a body weight of more than 50 kilograms (kg)

Exclusion Criteria:

* Have participated within the last 3 months in a clinical trial involving an investigational product
* Have known allergies to glucagon-like peptide-1 (GLP-1) analogs, or any components of the formulation, or history of significant atopy
* Have an abnormality in the 12-lead electrocardiogram (ECG) at screening and/or Day -1
* Have undergone any form of bariatric surgery
* Have obvious clinical signs or symptoms of liver disease, acute or chronic hepatitis
* Have a history of acute or chronic pancreatitis or elevation in serum lipase and/or amylase
* Show evidence of human immunodeficiency virus (HIV) or Hepatitis B or C
* Have used or intend to use medications that promote weight loss
* Have donated blood of more than 500 milliliter (mL) within the last month
* Currently smoke more than 10 cigarettes per day

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2016-12-05 (Actual); Primary Completion 2017-07-14 (Actual); Study Completion 2017-07-14 (Actual)

PRIMARY OUTCOMES:
Number of Participants with One or More Serious Adverse Event(s) (SAEs) considered by the Investigator to be Related to Study Drug Administration | Baseline to Study Completion (approximately 16 weeks)

SECONDARY OUTCOMES:
Pharmacokinetics (PK): Area Under the Concentration Curve (AUC) of LY3305677 | Day 1 Pre-dose through Day 85
Pharmacokinetics (PK): Maximum Drug Concentration (Cmax) of LY3305677 | Day 1 Pre-dose through Day 85

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST) or speak with your personal physician., Leeds, United Kingdom